CLINICAL TRIAL: NCT06241768
Title: Feasibility of a Cloud-based Digital Health Navigation Program for Colorectal Cancer Screening
Brief Title: Feasibility of a Colorectal Cancer Screening Web App in Primary Care Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Digital Health Navigation Solutions, Inc (Industry)
Collaborators: Wake Forest University Health Sciences (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 93476; R42CA275665 (NIH)
Record Dates: First submitted 2024-01-28; First posted 2024-02-05 (Actual); Results first posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Colorectal Cancer Screening
Keywords: colorectal cancer screening; pragmatic clinical trial; randomized clinical trial; digital health; feasibility study

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Text message 1 (Experimental): Version 1 of the text message invitation to use the cloud-based colorectal cancer screening program
  Interventions: Other: mPATH-CRC Web app
- Text message 2 (Experimental): Version 2 of the text message invitation to use the cloud-based colorectal cancer screening program
  Interventions: Other: mPATH-CRC Web app
- Text message 3 (Experimental): Version 3 of the text message invitation to use the cloud-based colorectal cancer screening program
  Interventions: Other: mPATH-CRC Web app
- Text message 4 (Experimental): Version 4 of the text message invitation to use the cloud-based colorectal cancer screening program
  Interventions: Other: mPATH-CRC Web app

INTERVENTIONS:
Other: mPATH-CRC Web app — Cloud-based web application that informs individuals of colorectal cancer screening and helps them receive screening

SUMMARY:
The goal of this clinical trial is to test the feasibility of a web app about colorectal cancer screening in patients with an upcoming primary care appointment. The main questions it aims to answer are:

* Among patients who use the web app, what proportion will request a colorectal cancer screening test via the program?
* How many patients will respond to a text message intervention to use the web app?

Participants will receive a text message informing them of the value of colorectal cancer screening, and inviting them to click a hyperlink to learn more. The hyperlink will take participants to the web app. The web app: 1) asks questions and use algorithms to determine if routine colorectal cancer screening is needed, and 2) if screening is indicated, shows a brief educational video about colorectal cancer screening and allows participants to request a screening test via the program.

Researchers will compare four different versions of the text message invitation to see if some messages result in higher program completion rates than others.

ELIGIBILITY:
Inclusion Criteria:

* Have a phone number listed in the electronic health record
* Language preference of English in the electronic health record
* Have a scheduled primary care appointment within the next 15 days

Exclusion Criteria:

* Prior diagnosis of colorectal cancer
* Prior diagnosis of inflammatory bowel disease
* Have a record in the electronic health record of completing a colonoscopy within the last 10 years, a FIT-DNA test within the last 3 years, or a fecal immunochemical test (FIT) within the last 1 year
* Have an electronic Charlson Comorbidity Index > 2

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 921 (Actual)
Dates: Start 2024-02-05 (Actual); Primary Completion 2024-03-26 (Actual); Study Completion 2024-03-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Miller, MD, MS, Principal Investigator — Digital Health Navigation Solutions, Inc
Locations (1):
- Atrium Health Wake Forest Baptist, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators will share the data dictionary and de-identified individual participant data that underlie our published results with researchers who provide a methodologically sound proposal. Use of the data will be limited to achieve the aims in their submitted proposal. To gain access, data requestors will need to sign a data access agreement.
Supporting Information: SAP
Time Frame: Individual participant data (IPD) and supporting information will be available beginning 6 months and ending 36 months following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal will be provided the data dictionary and deidentified participant data that underlie published study results. Use of the data will be limited to achieve the aims in their submitted proposal. To gain access, data requestors will need to sign a data access agreement. Researchers desiring IPD access should email requests to the study PI, Dr. David Miller (dave@mpathhealth.com).
URL: https://www.mpathhealth.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Text Message 1 | Text Message 2 | Text Message 3 | Text Message 4
Started | 232 | 230 | 229 | 230
Confirmed Eligible for CRC Screening | 29 | 35 | 34 | 37
Completed | 232 | 230 | 229 | 230
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Text Message 1 | Text Message 2 | Text Message 3 | Text Message 4 | Total
Number analyzed (Participants) | 232 | 230 | 229 | 230 | 921
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 191 | 180 | 177 | 182 | 730
  >=65 years | 41 | 50 | 52 | 48 | 191
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 134 | 142 | 137 | 138 | 551
  Male | 98 | 88 | 92 | 92 | 370
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 8 | 11 | 10 | 38
  Not Hispanic or Latino | 223 | 222 | 218 | 220 | 883
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 3 | 0 | 5
  Asian | 6 | 4 | 5 | 4 | 19
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 100 | 95 | 97 | 96 | 388
  White | 117 | 113 | 112 | 113 | 455
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 8 | 17 | 12 | 17 | 54
Region of Enrollment [Number; unit: participants]
  United States | 232 | 230 | 229 | 230 | 921

OUTCOME MEASURES:

1. Primary Outcome: Number (and Proportion) of Participants Who Request a Colorectal Cancer (CRC) Screening Test
Description: Number (and proportion) of participants who are confirmed eligible for CRC screening and request a CRC screening test within the mPATH-CRC Web App
Time Frame: 28 days
Population: Patients who used the mPATH-CRC Web App and were confirmed eligible for average-risk colorectal cancer screening
Measure: Count of Participants; unit: Participants
Arm/Group | Text Message 1 | Text Message 2 | Text Message 3 | Text Message 4
Number analyzed (Participants) | 29 | 35 | 34 | 37
Participants | 16 | 17 | 22 | 19

2. Secondary Outcome: Number (and Proportion) of Participants Who Complete the mPATH-CRC Web App
Description: Number (and proportion) of participants who complete the CRC screening eligibility questions within 4 weeks of the initial invitation using the mPATH-CRC Web App
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Text Message 1 | Text Message 2 | Text Message 3 | Text Message 4
Number analyzed (Participants) | 232 | 230 | 229 | 230
Participants | 55 | 66 | 51 | 59

ADVERSE EVENTS:
Time Frame: No adverse events were collected systematically for this study. The study intervention was a digital health program (a decision aid) for routine colorectal cancer screening as recommended by United States Preventive Services Task Force guidelines. Therefore, no adverse events were expected or collected.
Description: No adverse events were collected systematically for this study. The study intervention was a digital health program (a decision aid) for routine colorectal cancer screening as recommended by United States Preventive Services Task Force guidelines. Therefore, no adverse events were expected or collected.
Arm/Group | Text Message 1 | Text Message 2 | Text Message 3 | Text Message 4
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-01-25): https://cdn.clinicaltrials.gov/large-docs/68/NCT06241768/Prot_SAP_000.pdf